CLINICAL TRIAL: NCT02404428
Title: Effect of Sulforaphane on Prostate CAncer PrEvention-imagING Evaluation
Brief Title: Utilizing MRI to Study the Effect of Sulforaphane on Prostate Cancer
Acronym: ESCAPE-ING
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with recruitment
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: IFR02/2014
Record Dates: First submitted 2015-03-23; First posted 2015-03-31 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Prostate Cancer
Keywords: active surveillance; MRI; diet
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard broccoli soup (Active Comparator): one portion (300 g each) per week of a soup containing standard broccoli
  Interventions: Dietary Supplement: Standard broccoli soup
- beneforte extra broccoli soup (Experimental): one portion (300 g each) per week of a soup containing glucoraphanin-enriched broccoli named for the study 'Beneforte extra'
  Interventions: Dietary Supplement: Beneforte extra broccoli soup

INTERVENTIONS:
Dietary Supplement: Standard broccoli soup — 300g/week of standard broccoli soup consumed for a period of six months delivering standard level of glucoraphanin (sulforaphane precursor)
  Arms: standard broccoli soup
Dietary Supplement: Beneforte extra broccoli soup — 300g/week of beneforte extra broccoli soup consumed for a period of six months delivering enriched levels of glucoraphanin (sulforaphane precursor)
  Arms: beneforte extra broccoli soup

SUMMARY:
Prostate cancer is a major public health problem and there is a strong need of new preventive strategies based on drug and lifestyle interventions. It is now well-established that healthy eating patterns and increasing physical activity can prevent or delay prostate cancer progression. Intake of cruciferous vegetables (e.g. broccoli, cabbage, cauliflower, Brussels sprouts, kale) has been associated with decreased risk of prostate cancer progression; however the underlying biological mechanisms remain unknown. The investigators propose to undertake a pilot study on a group of men with early prostate cancer on active surveillance to determine whether a diet rich in broccoli will induce changes in tumor size and blood flow measured by conventional Magnetic Resonance Imaging (MRI) techniques. Men with early prostate cancer on active surveillance who have visible cancer lesions on MRI will be recruited onto this double-blinded randomized intervention and they will be asked to eat one portion of broccoli soup per week for 6 months. The investigators will test two varieties of broccoli (standard and 'Beneforte extra' broccoli) that are able to deliver two different levels of sulforaphane (SF), an active compound extensively studied for its potential anticancer properties. This study will involve MRI scans, blood and urine collection before and after a 6 month intervention period. This study design will not only allow us to observe diet-induced changes within the prostate but also at the systemic level. In addition, participant's lifestyle (habitual diet and physical activity) will be assessed by food diaries and exercise questionnaires.

This study has been funded by Biotechnology and Biological Sciences Research Council (BBSRC) and Prostate Cancer foundation (PCF).

DETAILED DESCRIPTION:
The study is a randomised double-blinded dietary intervention study. The study population will consist of men (n=20) aged 18-80 years with a BMI between 19.5 and 35 kg/m2 with low risk prostate cancer (prostate specific antigen [PSA] < 10ng/ml; Gleason grade 6; T category T1 or T2) or intermediate risk prostate cancer patients (PSA 10-20ng/ml; Gleason 7 (including selected 4+3 cases that will not be advised for radical prostatectomy; T category T1 or T2) who have visible lesions on MRI and have already decided to take up active surveillance/monitoring. The investigators chose these inclusion criteria because they reflect the population of men on active surveillance that the investigators are currently recruiting in the ESCAPE study (Effect of Sulforaphane on Prostate CAncer PrEvention; ClinicalTrials.gov Identifier: NCT01950143) via the Norfolk and Norwich University Hospital. Volunteers recruited onto this study will be randomly allocated to one of two arms in which they will be required to consume one portion of broccoli soup per week, delivering different levels of glucoraphanin (SF precursor) in each study arm. This will be part of their normal diet for 6 months. The two soups will contain standard broccoli (i), or glucoraphanin-enriched broccoli named for the study 'Beneforte extra' (ii). The study will involve MRI monitoring at baseline and after 6 months. In addition the investigators will collect blood and urine samples at baseline and after 6 months. The volunteers' habitual diet and physical activity will also be assessed during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Suitable for and have chosen AS as management for localised prostate cancer
* MRI visible detected lesion ≥0.5 cm in the axial plane, corresponding to the biopsy confirmed region of prostate cancer
* No contraindication to MR scanning
* Aged 18-80 years
* BMI between 19.5 and 35 kg/m2
* Smokers and non-smokers

Exclusion Criteria:

* 5α-reductase inhibitors or testosterone replacement medicines
* warfarin
* surgically implanted pelvic metalwork
* pacemakers or other implanted electronic devices not compatible with MRI
* contra-indications to gadolinium-based contrast agents (including patients with abnormal renal function)
* Glomerular Filtration Rate (GFR) <60 ml/min
* claustrophobia
* allergies to any of the ingredients of the broccoli soups
* dietary supplements or herbal remedies which may affect the study outcome - unless the volunteer is willing to discontinue taking them for 1 month prior to starting study
* parallel participation in another research project that involves dietary intervention

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
tumor size/blood flow | 6 months
  change in prostate tumor/blood flow size determined by MRI methods within the prostate gland

SECONDARY OUTCOMES:
choline + creatine/citrate ratio | 6 months
  concentration of metabolites (choline + creatine/citrate ratio) in the prostate tissue determined by using MR spectroscopy
citrate levels | 6 months
  concentration of citrate and associated metabolites in body fluids (blood, urine)
PSA levels | 6 months
  plasma levels of prostate-specific antigen (PSA) and other blood markers
GSTM1 genotype | 6 months
  Glutathione S-transferase Mu 1 (GSTM1) genotype or other relevant genotypes on mediating metabolite changes by diet

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mithen, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust_Addenbrooke's Hospital, Cambridge, United Kingdom